CLINICAL TRIAL: NCT02301936
Title: An Open-Label Study of Ledipasvir/Sofosbuvir Fixed-Dose Combination for 12 or 24 Weeks in Genotype 1 or 4 HCV Infected Subjects With Sickle Cell Disease
Brief Title: Ledipasvir/Sofosbuvir Fixed-Dose Combination for 12 or 24 Weeks in Genotype 1 or 4 HCV Infected Adults With Sickle Cell Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-1405
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2017-04

CONDITIONS: Hepatitis C Virus Infection
Keywords: Sickle Cell Disease; Gilead; Hepatitis C
MeSH Terms: conditions — Hepatitis C; Anemia, Sickle Cell | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LDV/SOF 12 weeks (Experimental): Treatment-naive or treatment-experienced participants without cirrhosis will receive LDV/SOF for 12 weeks.
  Interventions: Drug: LDV/SOF
- LDV/SOF 24 weeks (Experimental): Treatment-experienced participants with cirrhosis will receive LDV/SOF for 24 weeks.
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: LDV/SOF — 90/400 mg fixed dose combination (FDC) tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977

SUMMARY:
The primary objectives of this study are to evaluate the antiviral efficacy, safety, and tolerability of ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) administered for 12 or 24 weeks in adults with genotype 1 or 4 hepatitis C virus (HCV) infection with sickle cell disease (SCD).

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic genotype 1 or 4 infected patients with sickle cell disease
* HCV RNA ≥ 1,000 IU/mL at screening
* Cirrhosis determination by transient elastography
* Screening laboratory values within defined thresholds
* Use of two effective contraception methods if female of childbearing potential or sexually active male

Key Exclusion Criteria:

* Pregnant or nursing female
* Co-infection with HIV or hepatitis B virus (HBV)
* Current or prior history of clinical hepatic decompensation
* Hepatocellular carcinoma (HCC) or other malignancy (with exception of certain resolved skin cancers)
* History of clinically significant illness or any other medical disorder that may interfere with treatment, assessment or compliance with the protocol

Note: Other protocol defined inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2016-04-18 (Actual); Study Completion 2016-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (1):
- Lutherville, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 1 study site in the United States. The first participant was screened on 02 March 2015. The last study visit occurred on 18 April 2016.
Groups:
- LDV/SOF 12 Weeks: Treatment-naive or treatment-experienced participants without cirrhosis received ledipasvir/sofosbuvir (Harvoni®; LDV/SOF) 90/400 mg fixed dose combination (FDC) tablet once daily for 12 weeks
- LDV/SOF 24 Weeks: Treatment-experienced participants with cirrhosis received LDV/SOF 90/400 mg FDC tablet once daily for 24 weeks.
Period: Overall Study
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks
Started | 9 | 1
Completed | 8 | 1
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who took at least 1 dose of study drug.
Groups:
- LDV/SOF 12 Weeks: Treatment-naive or treatment-experienced participants without cirrhosis received LDV/SOF 90/400 mg FDC tablet once daily for 12 weeks
- Total: Total of all reporting groups
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks | Total
Number analyzed (Participants) | 9 | 1 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43 (14.9) | 44 (NA) — This treatment group had 1 participant only so standard deviation (SD) is not applicable. | 43 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 6 | 0 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 9 | 1 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 9 | 1 | 10
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 1 | 0 | 1
    CT | 2 | 1 | 3
    TT | 6 | 0 | 6
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 5.8 (0.74) | 6.2 (NA) — This treatment group had 1 participant only so SD is not applicable. | 5.8 (0.71)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 6 | 0 | 6
  ≥ 800,000 IU/mL | 3 | 1 | 4
HCV genotype [Count of Participants; unit: Participants]
  Genotype 1a | 5 | 1 | 6
  Genotype 1b | 1 | 0 | 1
  Genotype 4a/4c/4d | 1 | 0 | 1
  Genotype 4f | 1 | 0 | 1
  Genotype 4h | 1 | 0 | 1
Cirrhosis status [Count of Participants; unit: Participants]
  Absence | 9 | 0 | 9
  Presence | 0 | 1 | 1
Prior HCV Treatment Experience With Cirrhosis [Count of Participants; unit: Participants]
  Treatment-Naive (Non-cirrhosis) | 7 | 0 | 7
  Treatment-Experienced (Non-cirrhosis) | 2 | 0 | 2
  Treatment-Experienced (Cirrhosis) | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ) 12 weeks following the last dose of study drug.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who took at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks
Number analyzed (Participants) | 9 | 1
percentage of participants | 88.9 | 100.0

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 24 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks
Number analyzed (Participants) | 9 | 1
percentage of participants | 0 | 0

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < the LLOQ 4 weeks following the last dose of study drug.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks
Number analyzed (Participants) | 9 | 1
percentage of participants | 88.9 | 100.0

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ on Treatment
Time Frame: Weeks 1, 2, 4, 8,12, 16, 20, and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks
Number analyzed (Participants) | 9 | 1
percentage of participants
  Week 1 | 33.3 | 0
  Week 2 | 66.7 | 0
  Week 4 | 88.9 | 100.0
  Week 8 | 88.9 | 100.0
  Week 12 | 100.0 | 100.0
  Week 16: number analyzed (Participants) | 0 | 1
  Week 16 |  | 100.0
  Week 20: number analyzed (Participants) | 0 | 1
  Week 20 |  | 100.0
  Week 24: number analyzed (Participants) | 0 | 1
  Week 24 |  | 100.0

5. Secondary Outcome: HCV RNA Change From Baseline
Time Frame: Up to 24 weeks
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks
Number analyzed (Participants) | 9 | 1
log10 IU/mL
  Change at Week 1: number analyzed (Participants) | 6 | 1
  Change at Week 1 | -4.20 (0.543) | -3.86 (NA) — This group had only 1 participant so SD is not applicable.
  Change at Week 2 | -3.86 (1.644) | -4.63 (NA) — This group had only 1 participant so SD is not applicable.
  Change at Week 4 | -3.98 (1.694) | -5.05 (NA) — This group had only 1 participant so SD is not applicable.
  Change at Week 8 | -4.47 (0.662) | -5.05 (NA) — This group had only 1 participant so SD is not applicable.
  Change at Week 12 | -4.61 (0.737) | -5.05 (NA) — This group had only 1 participant so SD is not applicable.
  Change at Week 16: number analyzed (Participants) | 0 | 1
  Change at Week 16 |  | -5.05 (NA) — This group had only 1 participant so SD is not applicable.
  Change at Week 20: number analyzed (Participants) | 0 | 1
  Change at Week 20 |  | -5.05 (NA) — This group had only 1 participant so SD is not applicable.
  Change at Week 24: number analyzed (Participants) | 0 | 1
  Change at Week 24 |  | -5.05 (NA) — This group had only 1 participant so SD is not applicable.

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as
  * On-treatment virologic failure
    * HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ, while on treatment,
    * > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment, HCV RNA persistently ≥ LLOQ through 8 weeks of treatment (ie nonresponse)
  * Relapse
    * HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available posttreatment measurement
Time Frame: Up to Posttreatment Week 12
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks
Number analyzed (Participants) | 9 | 1
percentage of participants | 11.1 | 0

7. Secondary Outcome: Change From Pretreatment Assessment in Health-related Quality of Life as Evaluated by Short Form (SF-36) Health Survey Scale- Physical Component Score
Description: The SF-36 Health Survey is a self-reporting, multi-item scale measuring 8 health concepts: 1) physical functioning, 2) role limitations due to physical health problems, 3) bodily pain, 4) general health, 5) vitality (energy/fatigue), 6) social functioning, 7) role limitations due to emotional problems and 8) mental health (psychological distress and psychological well-being). The first 6 concepts constitute the physical component summary. The total score is an average of the individual question scores, which are scaled 0-100 with lower scores representing more disability and higher scores representing less disability.
Time Frame: Weeks 4,12, 24, Posttreatment Weeks 4 and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks
Number analyzed (Participants) | 9 | 1
units on a scale
  Week 4 | 1.2 (6.66) | 8.5 (NA) — This group had only 1 participant so SD is not applicable.
  Week 12 | 2.7 (7.20) | 5.8 (NA) — This group had only 1 participant so SD is not applicable.
  Week 24: number analyzed (Participants) | 0 | 1
  Week 24 |  | 2.3 (NA) — This group had only 1 participant so SD is not applicable.
  Posttreatment Week 4: number analyzed (Participants) | 8 | 1
  Posttreatment Week 4 | 3.5 (8.26) | 0.1 (NA) — This group had only 1 participant so SD is not applicable.
  Posttreatment Week 12: number analyzed (Participants) | 8 | 1
  Posttreatment Week 12 | 0.7 (12.46) | 5.5 (NA) — This group had only 1 participant so SD is not applicable.

8. Secondary Outcome: Change From Pretreatment Assessment in Health-related Quality of Life as Evaluated by Short Form (SF-36) Health Survey Scale- Mental Component Score
Description: The SF-36 Health Survey is a self-reporting, multi-item scale measuring 8 health concepts: 1) physical functioning, 2) role limitations due to physical health problems, 3) bodily pain, 4) general health, 5) vitality (energy/fatigue), 6) social functioning, 7) role limitations due to emotional problems and 8) mental health (psychological distress and psychological well-being). The last 5 concepts constitute the mental component summary. The total score is an average of the individual question scores, which are scaled 0-100 with lower score representing more disability and higher scores representing less disability.
Time Frame: Weeks 4,12, 24, Posttreatment Weeks 4 and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks
Number analyzed (Participants) | 9 | 1
units on a scale
  Week 4 | 2.2 (8.88) | -4.7 (NA) — This group had only 1 participant so SD is not applicable.
  Week 12 | 3.2 (8.14) | -3.3 (NA) — This group had only 1 participant so SD is not applicable.
  Week 24: number analyzed (Participants) | 0 | 1
  Week 24 |  | -3.9 (NA) — This group had only 1 participant so SD is not applicable.
  Posttreatment Week 4: number analyzed (Participants) | 8 | 1
  Posttreatment Week 4 | 2.2 (9.69) | -4.6 (NA) — This group had only 1 participant so SD is not applicable.
  Posttreatment Week 12: number analyzed (Participants) | 8 | 1
  Posttreatment Week 12 | 2.4 (6.53) | -5.0 (NA) — This group had only 1 participant so SD is not applicable.

9. Secondary Outcome: Change From Pretreatment Assessment in Health-related Quality of Life as Evaluated by Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F)
Description: The FACIT-Fatigue score was measured using a 40-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. Participants scored each item on a 5-point scale from 0 (Not at all) to 4 (Very much). The FACIT-F total score was calculated by taking the sum of all 40 individual scores and ranged from 0-160, with higher scores indicating better quality of life.
Time Frame: Weeks 4,12, 24, Posttreatment Weeks 4 and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks
Number analyzed (Participants) | 9 | 1
units on a scale
  Week 4: number analyzed (Participants) | 8 | 1
  Week 4 | 4.6 (13.86) | -0.2 (NA) — This group had only 1 participant so SD is not applicable.
  Week 12: number analyzed (Participants) | 8 | 1
  Week 12 | 9.8 (17.15) | 14.5 (NA) — This group had only 1 participant so SD is not applicable.
  Week 24: number analyzed (Participants) | 0 | 1
  Week 24 |  | 11.7 (NA) — This group had only 1 participant so SD is not applicable.
  Posttreatment Week 4: number analyzed (Participants) | 7 | 1
  Posttreatment Week 4 | 13.0 (17.20) | 13.2 (NA) — This group had only 1 participant so SD is not applicable.
  Posttreatment Week 24: number analyzed (Participants) | 7 | 1
  Posttreatment Week 24 | 8.5 (6.32) | 5.0 (NA) — This group had only 1 participant so SD is not applicable.

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF 24 Weeks
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/1
Other Adverse Events (participants affected / at risk) | 6/9 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 12 Weeks (N=9) | LDV/SOF 24 Weeks (N=1)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 12 Weeks (N=9) | LDV/SOF 24 Weeks (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 | 0
Eye discharge (Eye disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 6 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years